CLINICAL TRIAL: NCT03716167
Title: Randomized Controlled Trial for Treatment of Pain and Assessment of Wound Healing in Chronic Venous Leg Ulcers
Brief Title: Randomized Controlled Trial for Treatment of Pain and Assessment of Wound Healing in Chronic Venous Leg Ulcers Using Near Infrared Laser Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00040491
Record Dates: First submitted 2018-10-19; First posted 2018-10-23 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Venous Leg Ulcer
Keywords: laser; ulcer; wound
MeSH Terms: conditions — Varicose Ulcer; Ulcer; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Laser Treatment (Experimental): Summus Laser treatment with infrared light
  Interventions: Device: Summus Laser
- Sham treatment (Sham Comparator): Sham Summus Laser treatment with no infrared light
  Interventions: Device: Summus Laser Sham

INTERVENTIONS:
Device: Summus Laser — infrared laser treatment
  Arms: Laser Treatment
Device: Summus Laser Sham — non-infrared light
  Arms: Sham treatment

SUMMARY:
The laser emits an infrared light that heats the skin and underlying tissues with the purpose of temporary relief of minor muscle and joint pain, as well as stiffness associated with arthritis. The laser also causes a temporary increase in blood flow. The purpose of this study is to evaluate whether laser therapy can provide pain relief and speed the healing of venous leg ulcers.

DETAILED DESCRIPTION:
The Summus Laser Cube is an FDA cleared light-emitting device for applying infrared to provide topical heating for the purpose of elevating tissue temperature for temporary relief of minor muscle and joint pain, muscle spasm, pain and stiffness associated with arthritis and promoting relaxation of the muscle tissue and to temporarily increase local blood circulation.

There will be a total of 20 subjects involved in this study. The study will only involve participants being treated at the Wake Forest University Health Sciences Wound Care Center. Ten participants will be randomized to the treatment arm and receive therapeutic laser therapy applied to the ulcer area. The other ten participants will receive a sham laser therapy, where the light emitted by the laser is visible, but not powerful enough to provide a therapeutic effect. During the first weekly visit, patients will have the wound debrided (dead or dying tissue will be removed),and the size of the ulcer measured and photographed. A wound dressing will be applied, followed by a compression wrap.

After one week patients will return to the Wound Care clinic and the size of the wound will be evaluated. If the wound has decreased by less than 30%,the patient will be randomized into the protocol. The patient will then have weekly visits, to include a survey, wound measurements, survey, photos,and laser treatments. The length of the study is a maximum of 17 weeks (less if the patient heals faster). The purpose of this study is to evaluate whether laser therapy can provide pain relief and speed the healing of venous leg ulcers.

ELIGIBILITY:
Inclusion Criteria:

* 18 yo or older
* Venous insufficiency documented on basis of Venous Insufficiency US or on basis of skin changes c/w stasis
* Ulcer location in area of stasis present on lower limb
* Ulcer surface greater or equal to 5 cm2 but no larger than 140 cm2 after the initial debridement
* Ankle brachial index (ABI) > 0.8
* Ulcer duration longer than 4 weeks
* Pain scale assessment per visual analog scale at, or above, 2 at initial visit for the study

Exclusion Criteria:

* Pregnant, nursing or child bearing potential
* Venous ablation past 6 weeks and duration of study
* Autoimmune disorder
* Immune suppressive meds, Including steroids
* Any other co-playing comorbidities into wound etiology (neuropathy with pressure reinjury or uncontrolled diabetes with Hb A1c > 9)
* Use of bioengineered products 30 days before and during the duration of study
* 15<BMI <50
* Use of oral or IV administered antibiotics within one week prior to randomization
* Having tattoos in the region of skin above or adjacent to the ulcer where laser light might be applied.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-07-27 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Pain measured by survey | up to 17 weeks
  Survey of 0-10, with 0 being no pain and 10 being the worst pain imaginable

SECONDARY OUTCOMES:
Venous Ulcer rate of healing | up to 17 weeks
  healing rate to denote the length of time the patient has a wound
size of venous ulcer | up to 17 weeks
  wound measured length x width x depth
Infectious complications | up to 17 weeks
  Number of events of infectious complications
Wound aspect | up to 17 weeks
  % of granulation tissue
Quality of Life Questionnaire | up to 17 weeks
  Quality of life questions, 0 no trouble or 5 severe trouble

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Molnar, MD, Principal Investigator — WFUHS
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No